CLINICAL TRIAL: NCT01050959
Title: Compassionate Use Study of the Bion for Occipital Nerve Stimulation for Treatment of Chronic Headaches
Brief Title: Bion Occipital Nerve Stimulation (ONS) Compassionate Use Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4005; G030225/S022 (Other: FDA)
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2013-11

CONDITIONS: Chronic, Medically Refractory Headache
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: bion

SUMMARY:
The purpose of this compassionate use study is to provide clinical and technical support of the Bion® microstimulator system to the subjects who have decided to keep the system for relief of headache symptoms that have not responded to medical treatment. These study subjects were enrolled and implanted with the Bion® system during a previous clinical investigation of the Bion® for occipital nerve stimulation (ONS) in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Subject participated in a prior clinical feasibility study of the Bion for occipital nerve stimulation in the treatment of chronic headaches (IDE G030225) and remained implanted with the Bion system.
* Subject elects to enroll in this compassionate use study and provides written informed consent.
* Subject understands the type and duration of clinical, technical or product support provided in the study.
* Subject is willing to comply with protocol-required activities.

Exclusion Criteria:

* Subject is currently participating or intends to participate in another investigational drug or device clinical trial for chronic headaches during the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who were enrolled and implanted with the Bion® system during a prior feasibility clinical investigation of the device for occipital nerve stimulation (ONS) in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Provision of one year of clinical and technical support
  This is a compassionate use study. There are no primary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Chair — Boston Scientific Neuromodulation Corporation
Locations (2):
- United States (2):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan